CLINICAL TRIAL: NCT04576754
Title: Postpartum Depression Pivotal Test: Randomized Clinical Trial of WB001
Brief Title: Pivotal Test: WB001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woebot Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Woebot Labs Inc. - 0030
Record Dates: First submitted 2020-09-22; First posted 2020-10-06 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Models, Educational

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WB001 (Experimental)
  Interventions: Device: WB001
- Comparison Condition (Sham Comparator)
  Interventions: Device: Educational

INTERVENTIONS:
Device: WB001 — The WB001 treatment consists of PPD-specific psychoeducational lessons and CBT-specific skills or tools. The lessons teach PPD-specific information to normalize and contextualize postpartum experiences, as well as provide information on effective mood management and mental health promotion in the context of having recently given birth. Patients complete up to 30 psychoeducational lessons. In addition, patients access and apply core CBT-based tools upon endorsing a negative mood. These tools are core to CBT and are considered transdiagnostic. Examples include thought challenging, behavioral activation, mindfulness, and self-care.
  Arms: WB001
Device: Educational — The Comparison Condition provides educational only material about various mental and physical topics, delivered in an interactive smartphone application that is accessible anytime of day.
  Arms: Comparison Condition

SUMMARY:
The purpose of the present randomized controlled study is to investigate if there is a difference in postpartum depression symptoms among participants assigned to :

1. an automated conversational agent based on the most researched and scientifically validated psychotherapies, primarily Cognitive Behavioral Therapy (CBT), and accessible via an iOS and Android application, or to
2. a comparison condition without CBT and conversation, though still delivered in an interactive smartphone application that is accessible anytime of day.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years who had onset of a major depressive episode within the third trimester of pregnancy or within 4 weeks following delivery as measured by the MINI (Mini International Neuropsychiatric Interview).
* Current mild-moderate depression as measured by the HAM-D (HAM-D score>13 and <24)
* Women were </= to 6 months postpartum at the time of screening
* Owns a smartphone (Anrdroid or iOS smartphone with a recent, supported operating system)
* Available and committed to engage with the program and complete assessments for a 3-month duration
* Able to read and write in English
* U.S. resident

Exclusion Criteria:

* HAM-D score ≥ 24 (severe depression)
* Active psychosis
* Suicidal attempt or ideation with a plan and intent to harm oneself during the current episode of PPD
* History of (a) drug and/or alcohol abuse within the past 12 months (determined by self-report)
* Current pregnancy or plans to become pregnant within the next 4 months
* Fetal demise within the past 24 months
* Previous Woebot user

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale for Depression (HAMD) | Post-treatment at 8 weeks
  The HAMD is a 17-item, clinician rated measure of depression. Each item is scored from 0 to 2 and assesses the following criteria: insomnia, somatic symptoms, genital symptoms, loss of weight, and insight. The total score is calculated as a sum and ranges from 0 to 52, with higher scores indicating a greater degree of depression. The HAMD is commonly used for diagnostic purposes in research; structured clinical interviews such as this are recommended to actually diagnose clinical depression. It will be the primary outcome measure.

SECONDARY OUTCOMES:
Clinical Characteristic Questions | Baseline, Post-treatment at 8 weeks
  Questions assessing current and previous therapy, medication and diagnoses.
The Edinburgh Postnatal Depression Scale (EPDS) | Baseline, Mid-Treatment at 4 weeks, Post-treatment at 8 weeks, 1-Month Follow-up at 12 weeks
  The Edinburgh Postnatal Depression Scale (EPDS) is a validated screening for depressive symptomatology among women who have recently given birth. The instrument is recommended by the American College of Obstetricians and Gynecologists for postnatal depression screening for all postpartum individuals. It has 10 items that are scored on a 0-3 basis. For the purpose of this study item number 10 that inquires about suicidal ideation, was omitted. A total EPDS score will be utilized. A total score of 10 indicates possible depression and the maximum achievable is 30.
The Patient Health Questionnaire (PHQ-8) | Baseline, Mid-Treatment at 4 weeks, Post-treatment at 8 weeks, 1-Month Follow-up at 12 weeks
  The 8-item PHQ is an abbreviated version of the PHQ-9, will be used to assess mood and anxiety symptoms respectively. The PHQ-9 is a widely used self-report measure, with demonstrated reliability and sensitivity to clinical change. The PHQ-8 excludes an item assessing suicidality.
Generalized Anxiety Disorder 2-item scale (GAD-2) | Baseline, Mid-Treatment at 4 weeks, Post-treatment at 8 weeks, 1-Month Follow-up at 12 weeks
  The Generalized Anxiety Disorder 2-item scale (GAD-2) is a 2-item version of the GAD-7, a brief self-report tool to assess the frequency and severity of anxious thoughts and behaviors over the past 2 weeks. The correlation coefficient between the two measures was r=.75.
The Mother-to-Infant Bonding Scale (MIB) | Baseline, Mid-Treatment at 4 weeks, Post-treatment at 8 weeks, 1-Month Follow-up at 12 weeks
  The MIB consists of 8 one-word items describing an emotional response, such as ''loving'' or ''disappointed." Mothers rate the degree they feel the emotional response with their infant using a 4-point Likert scale from very much=0 to not at all=3. Five items describe negative emotional responses and are reverse scored. Total scores can range from 0 to 24, with lower scores indicating good bonding. Mother-infant bonding has been shown to be positively correlated with postpartum depression scores, where lower MIB are associated with lower depression scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) | Change from Baseline to Mid-Treatment at 4 weeks; Change from Baseline to Post-treatment at 8 weeks; Change from Baseline from12 weeks
  The PROMIS is a measure that evaluates and monitors physical, mental, and social health in adults and/or children. It can be used with the general population as well as with those living with chronic conditions. Each question has five response options ranging in value from 1-5. The total score is calculated by summing all items. Higher scores equal more of the concept being measured (e.g., more Fatigue, more Physical Function).
The Mental Health Self-Efficacy Scale (MHSES) | Baseline, Mid-Treatment at 4 weeks, Post-treatment at 8 weeks, 1-Month Follow-up at 12 weeks
  The MHSES was developed following Bandura's guidelines for constructing self-efficacy scales24. The six items assess confidence in managing stress, depression and anxiety, and are scored on a 10 point Likert scale (from 1, not at all confident to 10, very confident). Ratings across the 6 items are summed for an overall measure of MHSE (range 10 to 60), with higher scores indicating more self-efficacy. This measure is included as a way to capture an individual's confidence that they can successfully manage their mental health concerns.
The Client Satisfaction Questionnaire (CSQ-8) | Post-treatment at 8 weeks
  The CSQ-8 is an 8-item measure used to assess client's satisfaction with treatment on a 4-point scale (1= "very dissatisfied" to 4= "very satisfied") [15, 22] will be utilized starting at week 2 and continuing biweekly thereafter. Example questions include, "how would you rate the quality of service you received?" and "did you get the kind of service you wanted?" Total sums range from 8-32, with high scores indicating greater satisfaction with Woebot. The CSQ-8 has been widely disseminated and considered both valid and reliable (α ranges= .83-.93).

CONTACTS AND LOCATIONS:
Locations (1):
- Woebot Labs Inc, San Francisco, California, United States